CLINICAL TRIAL: NCT00500487
Title: Therapeutic Schools: Affect Management and HIV Prevention
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01MH066641 (NIH); R01MH066641 (NIH)
Record Dates: First submitted 2007-07-11; First posted 2007-07-12 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2009-10

CONDITIONS: HIV Infections
Keywords: HIV prevention; HIV seronegativity
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental)
  Interventions: Behavioral: Affect Management
- 2 (Active Comparator)
  Interventions: Behavioral: HIV Prevention Skills
- 3 (Active Comparator)
  Interventions: Behavioral: General Health Promotion

INTERVENTIONS:
Behavioral: Affect Management — 12-session group intervention including affect management training as well as sexual health skills training.
  Arms: 1
Behavioral: HIV Prevention Skills — 12-session group intervention including sexual health skills training.
  Arms: 2
Behavioral: General Health Promotion — 12-session group intervention including health information on a variety of health topics.
  Arms: 3

SUMMARY:
Adolescents are at risk for HIV because of sexual and drug behavior intiated during this developmental period. Those with psychological distress are less likely than their peers to benefit from frequently used skills-based interventions. It appears that emotional lability during sexual situations disrupts skills learned. This project will implement and evaluate interventions for adolescents with psychiatric disorders who are in therapeutic school settings. Affect management and skills-based interventions will be compared to a didactic standard of care condition to determine which intervention best reduces risk behavior among adolescents with psychiatric disorders in therapeutic school settings.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent attending therapeutic school

Exclusion Criteria:

* Adolescent is HIV positive
* Adolescent is developmentally delayed
* Adolescent is pregnant
* Adolescent has a history of sexual crime

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 420 (Estimated)
Dates: Start 2003-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Adolescent-reported condom use | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Larry K Brown, MD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Brown LK, Whiteley L, Houck CD, Craker LK, Lowery A, Beausoleil N, Donenberg G. The Role of Affect Management for HIV Risk Reduction for Youth in Alternative Schools. J Am Acad Child Adolesc Psychiatry. 2017 Jun;56(6):524-531. doi: 10.1016/j.jaac.2017.03.010. Epub 2017 Mar 31. PMID 28545758